CLINICAL TRIAL: NCT05815680
Title: A Study to Evaluate the Drug-drug Interactions (DDIs) of IBI362 With Metformin, Warfarin, Atorvastatin, Digoxin in Overweight or Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIBI362D101
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Overweight Subjects; Obese Subjects
MeSH Terms: interventions — Metformin; Digoxin; mazdutide; Warfarin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warfarin+atorvastatin+IBI362 (Experimental)
  Interventions: Drug: IBI362; Drug: warfarin; Drug: atorvastatin
- metformin+digoxin+IBI362 (Experimental)
  Interventions: Drug: metformin; Drug: digoxin; Drug: IBI362

INTERVENTIONS:
Drug: metformin — For oral administration, given as a single dose. The first dose is given before IBI362 treatment and the second dose is given at the end of IBI362 treatment.
  Arms: metformin+digoxin+IBI362
Drug: digoxin — For oral administration, given as a single dose. The first dose is given before IBI362 treatment and the second dose is given at the end of IBI362 treatment.
  Arms: metformin+digoxin+IBI362
Drug: IBI362 — Subjects will initiate treatment with 2 mg for the first four weeks followed by 4mg for four weeks and up to a dose of 6 mg for six weeks.
Drug: warfarin — For oral administration, given as a single dose. The first dose is given before IBI362 treatment and the second dose is given at the end of IBI362 treatment.
  Arms: warfarin+atorvastatin+IBI362
Drug: atorvastatin — For oral administration, given as a single dose. The first dose is given before IBI362 treatment and the second dose is given at the end of IBI362 treatment.
  Arms: warfarin+atorvastatin+IBI362

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate the influence of IBI362 on pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of warfarin, metformin, warfarin, atorvastatin, digoxin in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, age between 18 and 45 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 24 and 30 kg/m^2 (both inclusive) and weight≥50kg
* The subject has no birth plan and voluntarily takes effective contraceptive measures within 6 months after signing the informed consent form to the last medication

Exclusion Criteria:

* Cardiovascular, respiratory, hepatic, digestive (including digestive diseases that significantly affect gastric emptying or gastric motility, such as severe gastric spasticity or pyloric stenosis), endocrine (including but not limited to history of thyroid cancer or precancerous lesions), hematological and neurological disorders, or muscle degenerative disorders
* Drug or alcohol abuse
* Have dysphagia or any history of gastrointestinal diseases that affect drug absorption.
* Medical history or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
* Have a history of acute and chronic pancreatitis or serum amylase and/or lipase ≥ upper limit of normal value (Upper Limit of Normal value, ULN) at the time of screening.
* Those with a history of hypoglycemia.
* Previous or current mental illness.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed metformin plasma concentration at steady state | up to 116 days
Area under the metformin plasma concentration-time curve | up to 116 days
Maximum observed warfarin plasma concentration at steady state | up to 116 days
Area under the warfarin plasma concentration-time curve | up to 116 days
Maximum observed atorvastatin plasma concentration at steady state | up to 116 days
Area under the atorvastatin plasma concentration-time curve | up to 116 days
Maximum observed digoxin plasma concentration at steady state | up to 116 days
Area under the digoxin plasma concentration-time curve | up to 116 days

SECONDARY OUTCOMES:
Actual adverse events | up to 116 days
Terminal elimination half-life | up to 116 days
time to maximum plasma concentration of IBI362 | up to 116 days
Incremental area under the INR (international normalised ratio) -curve of warfarin | up to 116 days
Total apparent clearance of IBI362 | up to 116 days
Apparent volume of distribution of IBI362 | up to 116 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, Beijing Municipality, China